CLINICAL TRIAL: NCT01585064
Title: Optimization of Treatment With Adalimumab (HUMIRA): A Multi-center, Randomized, Single Blind, Controlled Clinical Trial
Brief Title: Optimization of Treatment With Adalimumab (Humira)
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Janet Pope, Prinicipal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: A06-216; HUM-05-081 (Other Grant/Funding Number: Abbott Laboratories Ltd.)
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis (RA); Anti-TNF therapy; Adalimumab; Disease activity; Treating to target
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- DAS28-IOMS: Physicians randomized to the DAS28-IOMS will treat patients according to a protocol aimed at achieving a DAS28 score under 2.4.
  Interventions: Other: DAS28-IOMS
- 0SJ-IOMS: Physicians randomized to the 0SJ-IOMS will treat patients according to a protocol aimed at attaining a count of zero swollen joint (28 joints evaluated).
  Interventions: Other: 0SJ-IOMS
- Routine Care (RC): Physicians randomized to the RC group will treat study patients as per routine care and according to their own judgment.
  Interventions: Other: Routine Care (RC)

INTERVENTIONS:
Other: DAS28-IOMS — Investigators randomized to DAS28-IOMS will be expected to adapt their therapeutic approaches in relation to the defined targets, i.e. to optimize adalimumab treatment according to individual patient's responses to treatment in order to achieve a DAS28 score of < 2.4.
  Groups: DAS28-IOMS
Other: 0SJ-IOMS — Investigators randomized to 0SJ-IOMS will be expected to adapt their therapeutic approaches in relation to the defined targets, i.e. to optimize adalimumab treatment according to individual patient's responses to treatment in order to achieve a swollen joint count of 0.
  Groups: 0SJ-IOMS
Other: Routine Care (RC) — Investigators randomized to RC will NOT be expected to adapt their therapeutic approaches to a pre-defined target. They will optimize adalimumab treatment according to individual patient's responses to treatment as per routine care and according to their own judgment.
  Groups: Routine Care (RC)

SUMMARY:
The purpose of this trial is to assess the effect of two Intensive Outpatient Management Strategies (IOMS) versus Routine Care (RC) on the outcomes of patients with Rheumatoid Arthritis (RA) that are treated with adalimumab.

This is a multi-center, randomized, controlled, parallel group, single (patient) blind trial. A total of 300 patients (100 per group) with RA will be recruited from approximately 40 sites across Canada.

DETAILED DESCRIPTION:
Background:

Rheumatoid arthritis (RA) is chronic systemic inflammatory disease often leading to damage and disability (Lee DM, et al.). RA is associated with a shorter life expectancy (Pincus T, et al.) and, if untreated, can lead to significantly lower quality of life and functional impairment (Bradley EM, et al.).

The concept of tight control, involving the treatment of patients to specified targets with close monitoring and treatment adjustment when necessary, has been trialed in early RA. Many targeted studies have demonstrated improved outcomes or faster target achievement in early RA.

The TICORA trial, which studied a group of patients who had active disease but who had not progressed to multiple DMARDs or biologic therapy, demonstrated that the usage of an intensive outpatient management strategy (IOMS) of RA improved clinical outcomes measures (Grigor C, et al.). Indeed, the results from this clinical trial have shown that strict control and intense follow up, which are based on titration of treatment in accordance to a standardized protocol, improved disease activity, physical function and quality of life of patients without additional cost.

The proposed study will evaluate the application of two types of IOMS. The first IOMS will consist of titration of treatments based on the attainment of a DAS28 score under 2.4 (DAS28-IOMS). The second IOMS will consist of titration of treatment based on the attainment of zero swollen joints (0SJ-IOMS) (28 joints evaluated). Investigators should aim at achieving those targets within a reasonable period of time, i.e. during the first six months of treatment with adalimumab. In addition, investigators should aim at attaining these targets within reasonable limits for each individual patient. The clinical impact of these two IOMS will be compared to that of routine care (RC).

The results of this study will have significant implications not only for the individual subjects but also from the societal perspective since it may enhance the overall real-life effectiveness of the treatments and will identify the best approach to maximize on the benefits of treatment with HUMIRA®.

Primary Objective:

In patients with RA that are initiated on treatment with adalimumab:

* The primary aim of the current study will be to assess the effect of two IOMS versus RC on the outcomes of patients with RA that are treated with adalimumab. The secondary aim will be to assess the differential effect of a DAS28-IOMS and a 0SJ-IOMS in this patient population.

Secondary Objectives:

In patients with RA that are initiated on treatment with adalimumab:

* To compare the therapeutic effectiveness of DAS28-IOMS, 0SJ-IOMS and RC as measured by the proportion of subjects achieving target scores of the DAS28.
* To compare the impact of DAS28-IOMS, 0SJ-IOMS and RC on patient subjective assessment of functional status as measured by the Health Assessment Questionnaire (HAQ).
* To compare the impact of DAS28-IOMS, 0SJ-IOMS and RC on patients' perception of their disease as evaluated by the Work Limitation Questionnaire (WLQ).
* To compare the impact of DAS28-IOMS, 0SJ-IOMS and RC on patients' satisfaction with care as evaluated by the change of patients' satisfaction measured on a Likert scale.
* To compare the therapeutic effectiveness of DAS28-IOMS, 0SJ-IOMS and RC as measured by the proportion of subjects achieving good or moderate European League against Rheumatism (EULAR) responses.
* To compare the impact of DAS28-IOMS, 0SJ-IOMS and RC on the frequency of serious adverse events or protocol-specified adverse events.

Tertiary Study Objectives:

In patients with RA that are initiated on treatment with adalimumab:

* To compare the therapeutic effectiveness of DAS28-IOMS, 0SJ-IOMS and RC as measured by the proportion of subjects achieving target scores of the CDAI and the SDAI.
* To describe the impact of individual components of the DAS28 on clinical decisions regarding patient management.
* To describe the impact of the CDAI on clinical decisions regarding patient management.
* To describe the impact of the SDAI on clinical decisions regarding patient management.
* To describe the impact of the HAQ on clinical decisions regarding patient management.
* To describe and compare the impact of a DAS28-IOMS, 0SJ-IOMS and RC on patients' compliance to treatment.
* To describe and compare the impact of a DAS28-IOMS, 0SJ-IOMS and RC on changes in concomitant anti-rheumatic medication use.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of rheumatoid arthritis
* Patient is > 18 years of age
* Patient is naïve to HUMIRA® (adalimumab) therapy.
* Patient has access to reimbursement for their standard of care.
* If female, patient is either: 1) not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or 2) of childbearing potential and practicing one of the following methods of birth control:

  * condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD)
  * contraceptives (oral or parenteral) for three months prior to enrollment in the study
  * a vasectomized partner
  * total abstinence from sexual intercourse
* If female and of childbearing potential, patient must have a negative serum pregnancy test performed at Screening.
* Patient is able to give written informed consent and to complete the survey requirements.

Exclusion Criteria:

* Patients had a history of cancer within the past 5 years other than a successfully treated basal cell carcinoma and/or localized carcinoma in situ of the cervix
* Patients with a history either of lymphoma or leukemia.
* Patients with a history of untreated active tuberculosis, or listeriosis, or other currently active infections suggestive of significant or profound immunosuppression, such as Pneumocystis carinii, aspergillosis or other systemic protozoal or fungal infections.
* Patients with a known positive HIV test.
* Patients with a known positive HepBsAg test.
* Patients with a persistent or severe infection(s) requiring hospitalization or treatment with iv antibiotics within 30 days, or oral antibiotics within 14 days, prior to enrollment.
* Female patients who are breast-feeding.
* Patients with clinically significant concurrent illness that in the investigator's judgment may influence the study outcomes (such as MS, moderate to severe CHF, etc,).
* Patients with any condition that would prevent participation or completion in this study including language limitation or possibility that the patient will not be available for the complete study period (18 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from approximately 40 sites across Canada. The study sample selection will be stratified in order to ensure adequate representation from all Canadian regions.
Sampling Method: Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in Disease Activity as measured by the DAS28 after 12 months of treatment | Baseline (0) and Month 12
  The change in DAS28 will be calculated as an absolute and percent value. The percent change in DAS28 will the calculated as [DAS28M12 - DAS28M0) / (DAS28M0} x 100% where: DAS28M12 is the DAS28 score at 12 months and - DAS28M0 is the DAS28 score at baseline.
  The DAS28 is a validated scale that measures disease activity in patients with rheumatic diseases. It is a composite scale that consists of the following: tender joint count, swollen joint count, ESR (mm/hr) and patient's global assessment of disease activity using a visual analog scale (VAS).

SECONDARY OUTCOMES:
Absolute and percent change in DAS28 | Baseline (0), Month 6, Month 12 and Month 18 (Study end)
  The DAS28 is a validated scale that measures disease activity in patients with rheumatic diseases. It is a composite scale that consists of the following: tender joint count, swollen joint count, ESR (mm/hr) and patient's global assessment of disease activity using a visual analog scale (VAS).
Absolute and percent change in the Health Assessment Questionnaire (HAQ) | Baseline (0), Month 6, Month 12 and Month 18 (Study end)
  The HAQ is a self-administered questionnaire to asses patient's health assessment and disability related to RA. The eight categories assessed by the HAQ are 1) dressing and grooming, 2) arising, 3) eating, 4) walking, 5) hygiene, 6) reach, 7) grip, and 8) common daily activities. For each of these categories, patients report the amount of difficulty they have in performing two or three specific activities. The HAQ score is the average of the worst score in each of the eight categories. The total score ranges from 0-3.
Absolute and percent change in individual components of the DAS28 | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  The DAS28 is a validated scale that measures disease activity in patients with rheumatic diseases. It is a composite scale that consists of the following: tender joint count, swollen joint count, ESR (mm/hr) and patient's global assessment of disease activity using a visual analog scale (VAS).
Percent achieving clinical remission defined as a DAS28 < 2.6 | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  The DAS28 is a validated scale that measures disease activity in patients with rheumatic diseases. It is a composite scale that consists of the following: tender joint count, swollen joint count, ESR (mm/hr) and patient's global assessment of disease activity using a visual analog scale (VAS).
Time to achieving clinical remission as measured by the DAS28 <2.6 | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  The DAS28 is a validated scale that measures disease activity in patients with rheumatic diseases. It is a composite scale that consists of the following: tender joint count, swollen joint count, ESR (mm/hr) and patient's global assessment of disease activity using a visual analog scale (VAS).
Percent achieving a DAS28 < 3.2 | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  The DAS28 is a validated scale that measures disease activity in patients with rheumatic diseases. It is a composite scale that consists of the following: tender joint count, swollen joint count, ESR (mm/hr) and patient's global assessment of disease activity using a visual analog scale (VAS).
Time to achieving a DAS28 <3.2 | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  The DAS28 is a validated scale that measures disease activity in patients with rheumatic diseases. It is a composite scale that consists of the following: tender joint count, swollen joint count, ESR (mm/hr) and patient's global assessment of disease activity using a visual analog scale (VAS).
Percent achieving a DAS28<2.4 | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  The DAS28 is a validated scale that measures disease activity in patients with rheumatic diseases. It is a composite scale that consists of the following: tender joint count, swollen joint count, ESR (mm/hr) and patient's global assessment of disease activity using a visual analog scale (VAS).
Time to achieving a DAS28<2.4 | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  The DAS28 is a validated scale that measures disease activity in patients with rheumatic diseases. It is a composite scale that consists of the following: tender joint count, swollen joint count, ESR (mm/hr) and patient's global assessment of disease activity using a visual analog scale (VAS).
Percentage achieving good or moderate European League Against Rheumatism (EULAR) responses | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  EULAR response criteria using DAS28 Score
Time to achieving good or moderate EULAR responses | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  EULAR response criteria using DAS28 Score
Patient Satisfaction with Care | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  A Likert scale will be used to evaluate the patient's satisfaction with care at each visit.
Absolute and percent change in the Work Limitations Questionnaire (WLQ) | Baseline (0), Month 6, Month 12 and Month 18 (Study end)
  The WLQ is used to measure the impairment in work related productivity, with reference to the previous two weeks.
Incidence of adverse events / serious adverse events | Baseline (0), Month 6, Month 12, Month 18 (Study End)
  All adverse events will be coded according to the MedDRA dictionary of terms and will be classified according to causal association to adalimumab (HUMIRA®). All events will be reported by body system using MedDRA preferred terms. The incidence rates of adverse events will be described as the proportion of subjects experiencing at least one event and as the number of events per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, MD MPH FRCPC, Principal Investigator — Lawson Health Research Institute, Western University
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

REFERENCES:
- [Background] Lee DM, Weinblatt ME. Rheumatoid arthritis. Lancet. 2001 Sep 15;358(9285):903-11. doi: 10.1016/S0140-6736(01)06075-5. PMID 11567728
- [Background] Pincus T, Callahan LF. Taking mortality in rheumatoid arthritis seriously--predictive markers, socioeconomic status and comorbidity. J Rheumatol. 1986 Oct;13(5):841-5. No abstract available. PMID 3820193
- [Background] Badley EM, Rasooly I, Webster GK. Relative importance of musculoskeletal disorders as a cause of chronic health problems, disability, and health care utilization: findings from the 1990 Ontario Health Survey. J Rheumatol. 1994 Mar;21(3):505-14. PMID 8006895
- [Background] Grigor C, Capell H, Stirling A, McMahon AD, Lock P, Vallance R, Kincaid W, Porter D. Effect of a treatment strategy of tight control for rheumatoid arthritis (the TICORA study): a single-blind randomised controlled trial. Lancet. 2004 Jul 17-23;364(9430):263-9. doi: 10.1016/S0140-6736(04)16676-2. PMID 15262104
- [Derived] Pope JE, Haraoui B, Rampakakis E, Psaradellis E, Thorne C, Sampalis JS; Optimization of Adalimumab Trial Investigators. Treating to a target in established active rheumatoid arthritis patients receiving a tumor necrosis factor inhibitor: results from a real-world cluster-randomized adalimumab trial. Arthritis Care Res (Hoboken). 2013 Sep;65(9):1401-9. doi: 10.1002/acr.22010. PMID 23509040
- [Derived] Pope J, Thorne JC, Haraoui BP, Psaradellis E, Sampalis J. Do patients with active RA have differences in disease activity and perceptions if anti-TNF naive versus anti-TNF experienced? Baseline results of the optimization of adalimumab trial. Med Sci Monit. 2012 Aug;18(8):PI17-20. doi: 10.12659/msm.883250. PMID 22847212